CLINICAL TRIAL: NCT07245134
Title: Virtual Reality Exposure Therapy in Patients With Obsessive-Compulsive Disorder: A Randomized Controlled Trial in Inpatients
Brief Title: Virtual Reality Exposure Therapy for Obsessive-Compulsive Disorder: A Randomized Controlled Trial in Inpatients
Acronym: OCD-VRET1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Principal Investigator, Iveta Fajnerová, Supervisor, National Institute of Mental Health, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU23-04-00402_Study1
Record Dates: First submitted 2025-09-25; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Obsessive-Compulsive Disorder; Virtual Reality Exposure Therapy; Virtual Reality Cognitive Training; Cognitive Behavior Therapy
Keywords: obsessive-compulsive disorder; VR exposure therapy; cognitive flexibility; Inpatient clinic
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Virtual Reality Exposure Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality exposure (Experimental): Participants complete 6-week CBT program with five 30-40-minute sessions of exposure administered via a virtual reality headset (once a week). The intervention involves exposure to various symptom provoking scenarios in the virtual house environment - "OCD house". Scenarios can be adjusted to distinct OCD dimensions: contamination/cleaning, fear-of-harm/checking, symmetry/ordering. Stimuli can be also freely combined across dimensions, so that the scenarios fit to individual needs.
  Interventions: Behavioral: Exposure Therapy (Virtual Reality)
- Cognitive flexibility training (Active Comparator): Control group attends 6-week CBT program with five sessions of 30-40 minutes of cognitive training via virtual reality headset using "VRcity" cognitive training games.
  Interventions: Behavioral: Cognitive flexibility training
- Standard CBT without additional VR treatment (Active Comparator): Control group completes the standard 6-week CBT program only, with no VR sessions.
  Interventions: Behavioral: Standard CBT program without VR interventions

INTERVENTIONS:
Behavioral: Exposure Therapy (Virtual Reality) — Virtual reality scenarios consists of exposures to OCD symptom provoking stimuli and response prevention (e.g. having dirty hands without washing them immediately) with the support of the therapist. The goal of VRET is sufficient reduction in anxiety and acceleration of progress in classical CBT.
  Arms: Virtual reality exposure
Behavioral: Cognitive flexibility training — Participants play series of various cognitive games previously developed in NIMH aimed at cognitive flexibility. Games are presented using immersive VR (HTC vive headset). The set includes for instance Go/No-go paradigm with a shooting range addressing inhibitory control, Flies - hit a fly game addressing set-shifting and Castle game addressing spatial memory and reversal learning.
  Arms: Cognitive flexibility training
Behavioral: Standard CBT program without VR interventions — Standart CBT program (performed in all groups). The program involves regular group and individual psychotherapy sessions 5 days per 6 weeks.
  Other Names: Cognitive Behavior Therapy
  Arms: Standard CBT without additional VR treatment

SUMMARY:
The aim of this study is to evaluate the efficacy of virtual reality exposure therapy (VRET) as a treatment for obsessive-compulsive disorder (OCD). Participants are randomly assigned to one of the following interventions: a) exposure condition - the group with a standard CBT program enriched with exposure therapy in VR (VRET), b) control condition 1 - the group with a standard CBT program enriched with VR cognitive training aimed at cognitive flexibility or c) control condition 2 - standard CBT program without any additional VR intervention. The treatment effect will be evaluated using pre/post assessments, as well as monitoring adherence to exposure and response prevention assignments.

DETAILED DESCRIPTION:
The virtual environment of so called "OCD house" is used as a tool for the intervention in the experimental group. Immersive VR glasses HTC Vive Pro are used to visualize the virtual environment.

During exposure therapy, relevant virtual stimuli can be freely combined involving common objects and situations in the home that may trigger OCD symptoms and hoarding behavior. Target stimuli (VR elements) are divided into several sets corresponding to OCD subtypes. During the session, the therapist can modify the level of difficulty via four standardized levels according to the individual needs of the clients.

The therapeutic application enables movement and direct interaction with stimuli in the environment of the virtual house and garden, thanks to a set of handhold controllers. Direct head and body rotations and small body movements are enabled by the VR headset. The psychotherapist can follow the patient actions and control the settings of the environment (e.g.selection of relevant stimuli, level of difficulty) using the computer and screen connected to the headset, and advise the patient where necessary. The level of difficulty is gradually increased during the progress of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD (F42) using currently valid DSM-V and ICD-11
* Fluent in Czech

Exclusion Criteria:

* Any other psychiatric, neurological and serious somatic illness
* Substance abuse
* Psychotropic medication (e.g. benzodiazepines) except antidepressants, antipsychotic medication and hypnotics.
* Contradictions to using a virtual reality (e.g., epilepsy, balance problems)
* Pregnancy
* Cardiostimulator and mental implants

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | Applied repeatedly: 1) At the baseline - Before the start of the first therapy session (S1), 2) Post-intervention - after the last session (S5) and 3) 2 months after the last session in the follow-up measurement (subjective Y-BOCS).
  The Y-BOCS is a 19-item scale assessing the severity of obsessive-compulsive symptoms. Raw score range from 0 to 40, where 0 = no symptoms and 40 = very severe symptoms with highly impaired daily functioning.
The Beck Depression Inventory (BDI) | Applied repeatedly for 5 weeks of the intervention (once per week) and 2 months after the last session in the follow-up measurement.
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Beck Anxiety Inventory (BAI) | Applied repeatedly for 5 weeks of the intervention (once per week) and 2 months after the last session in the follow-up measurement.
  BAI is an inventory of anxiety symptoms with 18 items rated on a 5-point Likert scale (0-4). Score range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Adherence to exposures | Immediately before each session (S1-S5) and 2 months after the last session in the follow-up measurement.
  Four questions aimed at gathering information about how patients managed to perform exposures during the past week and to what extent the skills acquired during the VR exposure therapy were useful.

SECONDARY OUTCOMES:
The Spielberger State-Trait Anxiety Inventory-X2 (STAI-X2) | 1) At the baseline - Before the start of the first therapy session (S1), 2) Post-intervention - after the last session (S5) and 3) 2 months after the last session in the follow-up measurement.
  The Spielberger State-Trait Anxiety Inventory-X2 (STAI-X2) is used to measure self-reported symptoms of trait anxiety with higher score indicating higher anxiety levels (score range 20-80).
Six-item State-Trait Anxiety Inventory (STAI-6) | Applied repeatedly during the intervention - twice during each of the 5 weekly sessions - Immediately Pre- and Post-Session (all sessions S1-S5)
  The 6-item short form of the Spielberger State-Trait Anxiety Inventory is used to measure self-reported symptoms of state anxiety with higher score indicating higher anxiety levels.
Subjective Units of Distress Scale (SUDS) | During In-Sessions: all sessions S1-S5
  The SUDS is a visual analog scale in which the participant rates his/her anxiety/discomfort based on a range between 1 (no anxiety/discomfort) and 10 (very severe anxiety/discomfort).
Anxiety Hierarchy | Baseline - Immediately before first (S1), posttreatment - after the last session (S5) + (Controlling for Baseline Score) and 2 months after the last session in the follow-up measurement.
  The patient is asked to develope a hierarchy of feared situations ranging from most-feared at the top to least-feared at the bottom. Then, he/she rates anticipated fear, anxiety or distress for each item (score 1-10, with higher score indicating higher anxiety) - according to how distressing they feel it would be to encounter that situation. The hierarchy is used to guide a process of VRET sessions.
Barratt Impusiveness Scale (BIS-11) | Immediately before the first (S1), after the last (S5) session and 2 months after the last session in the follow-up measurement.
  BIS is a 30-item scale used for self-assessment of impulsivity. Participants rate each item on a 4-point scale. Total score range from 30 to 120, where higher scores indicate higher impulsivity.
Cognitive Flexibility Inventory | Immediately before the first (S1), after the last (S5) session and 2 months after the last session in the follow-up measurement.
  CFI is self-report measure of the type of cognitive flexibility necessary for replace maladaptive thoughts with more balanced thinking. It has 20-items that participants evaluate on a 7-point Likert scale. The total score ranges from 20 to 140 and higher scores indicate more cognitive flexibility.

OTHER OUTCOMES:
The Igroup Presence Questionnaire (IPQ) | Immediately after second session (S2)
  The scale includes 3 subscales SP (spatial presence), INV (involvement) and REAL (experienced realism) with score range 0-7. Higher scores indication higher sense of presence. This measure might be positivelly associated with positive outcome.
Simulator Sickness Questionnaire (SSQ) | Immediately after second session (S2)
  The scale evaluates cybersickness symptoms in three subscales: nausea (N), oculomotor disturbance (O), disorientation (D). Total simulator sickness raw score 0-48 (adjusted total score 0-180). Higher scores on each scale indicate stronger perceptions of the underlying sickness symptoms and are therefore undesired. This measure might be negatively associated with positive outcome and sense of presence.

CONTACTS AND LOCATIONS:
Overall Officials: Iveta Fajnerová, Ph.D., Study Director — National Institute of Mental Health (NIMH); Pavla Stopková, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health, Klecany, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the publication of results, minimum of 5 years
Supporting Information: Study Protocol, SAP
Time Frame: Immediately after the publication of study results, at least for 5 years.
Access Criteria: The anonymized preprocessed behavioral data will be shared using an institutional open access or journal repository. Additional raw data access requests will be reviewed using an online form. Requestors will be required to sign a data access agreement.